CLINICAL TRIAL: NCT05658874
Title: A Multidisciplinary, Multimodal Bundled Care Approach to Chronic Pelvic Pain
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jocelyn Fitzgerald (Other)
Responsible Party: Sponsor-Investigator, Jocelyn Fitzgerald, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21060060
Record Dates: First submitted 2022-11-23; First posted 2022-12-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Therapeutics; Administration, Intravesical; Methenamine; Amitriptyline; Gabapentin

STUDY DESIGN:
Intervention Model Description: Single center, randomized pre-post intervention/prospective cohort study of usual Urogynecology care vs. multimodal, multidisciplinary care bundle (MMCB).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal care bundle (Experimental): Components of multimodal care bundle
  1. MD Evaluation
  2. On site pelvic floor physical therapy
  3. Behavioral health consult with appropriate psychiatric referrals/treatments
  4. Central sensitization/neurogenic pain:
     Amitriptyline 10-50mg Or Gabapentin (doses range from 100mg po tid to 600mg po tid)
  5. Urinary symptoms IC/PBS:
     Spasm: Overactive bladder medication chosen based on patient characteristics/insurance, dose may be increased as tolerated (Oxybutynin/Trospium/Detrol vs. Mirabegron)
  6. Microbiome: Methenamine
  7. Vaginal estrogen
     At least once within 12 weeks of initial visit:
  8. Operative cystoscopy
  9. Bladder instillations x 6 weeks (lidocaine, heparin, sodium bicarb, Kenalog, gentamicin)
  10. Pudendal/Levator and/or Obturator internus nerve block (120mg Kenalog and 0.25% Marcaine, total 23cc)
  Interventions: Drug: Multimodal Bundle Drugs; Procedure: Operative Cystoscopy; Behavioral: Behavioral health consultation/therapy; Other: Pelvic floor physical therapy; Drug: Bladder Instillation; Drug: Vaginal estrogen; Drug: Methenamine; Drug: Amitriptyline/Gabapentin
- Usual care (Active Comparator): IC/PBS treatments as directed by Urogynecology specialist
  Interventions: Other: Usual Urogynecologic care

INTERVENTIONS:
Drug: Multimodal Bundle Drugs — multimodal pain therapy
  Other Names: Overactive Bladder Medication( Trospium/Oxybutynin/Detrol vs. Mirabegron)
  Arms: Multimodal care bundle
Procedure: Operative Cystoscopy — Evaluate bladder and treat Hunner lesions with kenalog or fulguration as appropriate
  Arms: Multimodal care bundle
Behavioral: Behavioral health consultation/therapy — Patient to see behavioral health/psychiatric care
  Arms: Multimodal care bundle
Other: Pelvic floor physical therapy — Patient to have evaluation and treatment by a trained pelvic floor physical therapist
  Arms: Multimodal care bundle
Other: Usual Urogynecologic care — Usual care from practicing academic Urogynecologist
  Arms: Usual care
Drug: Bladder Instillation — Intravesical lidocaine, heparin, sodium bicarb, Kenalog, gentamicin
  Arms: Multimodal care bundle
Drug: Vaginal estrogen — Topical vaginal estradiol application
  Arms: Multimodal care bundle
Drug: Methenamine — UTI prevention/bladder therapeutic
  Arms: Multimodal care bundle
Drug: Amitriptyline/Gabapentin — Part of multimodal pain therapy
  Arms: Multimodal care bundle

SUMMARY:
The goal of this clinical trial is to compare two different treatment patterns in patients with chronic bladder pain. The main questions the investigators are seeking to answer is if bladder pain improves before and after treatment using a painful bladder scale. The participant will have 5 visits to evaluate your symptoms with questionnaires, at least one procedural visit, and must participate in physical therapy and some kind of behavioral health therapy. This study will assess participant response to a bundled-care approach to chronic bladder pain both pre-and post intervention as well as compared to a group of participants receiving typical care.

DETAILED DESCRIPTION:
Objectives:

The goals of this research program are to evaluate the patient-reported outcomes of a multimodal care bundle for patients presenting to a multidisciplinary chronic pelvic pain clinic compared to "usual care" in an Urogynecology clinic.

Primary Aim:

To compare pre and post intervention self-evaluation of pain and function scores in women with chronic pain syndromes with a primary finding of urinary/bladder pain symptoms with or without levator spasm who undergo multi-disciplinary, bundled care compared with usual care in a Urogynecology clinic setting.

Secondary Aims:

a) To identify and phenotype "non-responders" to a bundled approach to Interstitial Cystitis/Painful Bladder Syndrome/Chronic Pelvic Pain (IC/PBS/CPP).

Hypothesis: We hypothesize that a bundled, multidisciplinary care approach will significantly improve patient scores on validated outcomes questionnaires compared to usual care.

Methods:

All treatment plans, medications, and procedures recommended for patients involved in this study are within the current standards of care for IC/PBS/CPP, regardless of treatment arm and are known to be safe interventions.

Study Design: Single center, randomized pre-post intervention/prospective cohort study32 of usual FPMRS care vs. multimodal, multidisciplinary care bundle (MMCB).

Setting: Patients will be recruited from an outpatient Urogynecology clinic. They will subsequently be randomized to a Multidisciplinary chronic pelvic pain clinic at an alternate site vs. continuing usual outpatient care in Urogynecology as above.

ELIGIBILITY:
* Inclusion Criteria:
* Female patient 18 years of age or older
* diagnosis of Interstitial Cystitis/Painful Bladder Syndrome, scoring 6 points or higher on O'Leary Sant Questionnaire
* Exclusion Criteria:

Active pelvic or bladder infection within past 2 weeks

* contraindications to medications or intervention therapeutics
* inability to speak or read English
* pelvic floor interventional procedure including bladder instillations 4 weeks prior to study recruitment
* meets criteria for diagnostic laparoscopy
* internal referral (to reduce severity bias)

Note: patients are not excluded for currently taking any medication on the treatment list.

Patients can be treated for UTI during the study period.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
--O'Leary Sant Questionnaire (OLS), comprised of Interstitial Cystitis Symptom Index (ICSI) and Problem Index (ICPI), at 12 weeks from baseline MCID: 4 points for ICSI Change in O'Leary Sant Questionnaire Scores >4 points | 12 weeks
  Validated Questionnaire for evaluating Interstitial Cystitis. Scale range ICSI 0-20, ICPI 0-16, total 0-36. Higher score=worse pain. Improvement of 1-2 point is consider clinically significant.

SECONDARY OUTCOMES:
Healthcare encounters | 1 year
  Number of encounters with the UPMC healthcare system

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn J Fitzgerald, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No